CLINICAL TRIAL: NCT07185477
Title: A Single-arm Single-center Trial of Bridging GPRC5D/CD3 Bispecific Antibody Treatment With BCMA CAR-T Cell Therapy for Relapsed/Refractory Multiple Myeloma
Acronym: QLS32015
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025080; Qilu Pharmaceutical Co., Ltd. (Other Grant/Funding Number: Qilu Pharmaceutical Co., Ltd.)
Record Dates: First submitted 2025-09-05; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Relapsed/Refractory Multiple Myeloma (RRMM)
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QLS32015 (Experimental)
  Interventions: Biological: QLS32015

INTERVENTIONS:
Biological: QLS32015 — QLS32015 is a GPRC5D × CD3 bispecific antibody.

SUMMARY:
This study is a prospective, single-arm, multicenter trial designed to evaluate the hematologic response rate and safety of GPRC5D/CD3 bispecific antibody bridging therapy prior to CAR-T cell infusion in patients with relapsed/refractory multiple myeloma (RRMM).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary Participation: Ability to understand and voluntarily sign the informed consent form (ICF).
2. Age ≥18 years.
3. Confirmed symptomatic MM diagnosis per the Chinese Guidelines for Diagnosis and Management of Multiple Myeloma (2022 Revision).
4. Relapsed/Refractory MM (RRMM) meeting one of the following:

   Triple-class refractory RRMM: Resistant to ≥1 immunomodulatory drug (IMiD), ≥1 proteasome inhibitor (PI), and ≥1 anti-CD38 monoclonal antibody.

   Penta-drug refractory RRMM: Resistant to ≥2 IMiDs, ≥2 PIs, and ≥1 anti-CD38 antibody.

   Secondary plasma cell leukemia (sPCL):

   MM diagnosis per Chinese Guidelines (2022), plus Peripheral blood plasma cells ≥20% of leukocytes or absolute circulating plasma cells >2×10⁹/L.
5. Successful apheresis for CAR-T cell manufacturing.
6. ECOG performance status ≤3.
7. No active infections:

   HBV-DNA negative, HCV-RNA negative, HIV negative.
8. Liver function:

   Total bilirubin <1.5×ULN (<3×ULN for Gilbert's syndrome). AST/ALT <3×ULN.
9. Renal function: Calculated CrCl ≥30 mL/min (Cockcroft-Gault formula).
10. Baseline oxygen saturation >92% (room air).
11. Hematologic criteria (within 7 days of screening):

WBC ≥1.0×10⁹/L, ANC ≥1.0×10⁹/L, hemoglobin ≥70 g/L, and Platelets ≥75×10⁹/L (or ≥50×10⁹/L if bone marrow plasma cells ≥50%). Investigator discretion permitted for clinical justification. 12.Growth factor restrictions: 2-week washout required for erythropoietin, G-CSF, GM-CSF, or thrombopoietin agonists (e.g., eltrombopag).

13.Reproductive requirements: Non-childbearing women eligible; Childbearing potential women: Negative serum/urine pregnancy test (β-hCG) at screening.

14.Contraception: Males/females of reproductive potential must use effective contraception (per investigator judgment) during treatment and for ≥3 months post CAR-T infusion.

15.Sperm donation prohibition: Males must refrain from sperm donation from screening until 90 days post-treatment.

16.Compliance: Willing and able to complete study procedures and follow-up.

Exclusion Criteria:

1. Prior GPRC5D-targeted immunotherapy.
2. Investigator-assessed contraindications to GPRC5D×CD3 bispecific antibody therapy (e.g., severe cardiopulmonary diseases incompatible with treatment).
3. Grade >2 peripheral neuropathy or ≥grade 2 painful neuropathy at screening (regardless of current medication).
4. Known intolerance, hypersensitivity, or contraindication to GPRC5D×CD3 bispecific antibody components.
5. Initiation of bridging therapy for BCMA CAR-T cell treatment.
6. Unstable/active cardiovascular or cerebrovascular disease, including any of:

   1. Unstable angina, symptomatic myocardial ischemia, myocardial infarction, or coronary revascularization within 180 days prior to first dose.
   2. Uncontrolled hypertension (>140/90 mmHg with historical readings >180/100 mmHg within 6 months).
   3. Clinically significant uncontrolled arrhythmias (excluded: asymptomatic 1st-degree AV block or LAFB/RBBB).
   4. LVEF <40% by echocardiography.
   5. Stroke or intracranial hemorrhage within 12 months before screening.
   6. Pre-treatment severe thrombotic events.
7. Active HIV infection or seropositivity.
8. Active HBV/HCV infection:

   HBV: HBsAg(+) requires confirmed negative HBV-DNA PCR (allowed: if on antiviral therapy with confirmed suppression).

   HCV: HCV Ab(+) requires negative HCV-RNA PCR.
9. Pregnancy or lactation.
10. Active gastrointestinal disorders affecting swallowing or drug absorption.
11. Major surgery within 2 weeks pre-enrollment or planned during study (excluded: kyphoplasty/vertebroplasty; allowed: local anesthesia procedures).
12. Live vaccines within 4 weeks before first study dose.
13. Active psychiatric/medical conditions impairing compliance/consent capacity per investigator judgment.
14. Contraindications to required concomitant medications/supportive care.
15. Any condition interfering with study procedures.
16. Inability/unwillingness to comply with protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Minimum 2 years after infusion
  The proportion of subjects achieving stringent complete response (sCR), complete response (CR), very good partial response (VGPR), and partial response (PR) after treatment with QLS32015 injection
Safety and Tolerability | Minimum 2 years after infusion
  The incidence of treatment-emergent adverse events (TEAES)

SECONDARY OUTCOMES:
Time to Response (TTR) | Minimum 2 years after infusion
  Time from first BCMA×CD3 bispecific antibody infusion to first hematologic response，Depth of best hematologic response: The highest-level response achieved at any timepoint
Duration of Response (DOR) | Minimum 2 years after infusion
  Duration of response (DOR) was defined as the time from first documented hematologic response (≥ partial response [PR]) to disease progression or death due to progression, whichever occurred first
Overall Survival (OS) | Minimum 2 years after infusion
Progression-Free Survival (PFS) | Minimum 2 years after infusion

IPD SHARING:
Plan to Share IPD: No